CLINICAL TRIAL: NCT02977637
Title: The Use of Ferumoxytol (Feraheme) for Whole Body Magnetic Resonance Angiography in Hereditary Hemorrhagic Telangiectasia
Brief Title: MRA With Feraheme in HHT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Justin McWilliams, MD, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-001308
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: hht; hereditary; hemorrhagic; telangiectasia; feraheme
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Telangiectasis | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Feraheme group (Experimental): All patients enrolled in the study will receive Feraheme MRI/MRA to detect vascular malformations. Ferumoxytol in its standard concentration (510 mg in 17 cc) will be administered IV at 0.15-0.21 mg/kg prior to MRI/MRA.
  Interventions: Procedure: Feraheme MRI/MRA

INTERVENTIONS:
Procedure: Feraheme MRI/MRA
  Other Names: Ferumoxytol

SUMMARY:
Magnetic resonance (MR) imaging is performed with contrast agents to highlight the blood vessels and allow interpretation and diagnosis of blood vessel abnormalities. HHT (Hereditary Hemorrhagic Telangiectasia) is a disease of blood vessels, and can suffer fatal bleeding if abnormal blood vessels are not detected and treated early. Patients with HHT also require many imaging studies through their lifetimes for surveillance of blood vessels. Many HHT patients also have co-existing iron deficiency anemia from bleeding in their nose and gastrointestinal tract, and receive daily iron therapy.

Ferumoxytol is an alternative MR contrast agent, which is FDA (Food and Drug Administration) approved for the treatment of iron deficiency anemia. In addition, it is not associated with the risks to the kidneys of the other agents. The use of ferumoxytol for MR imaging may benefit the patients who do not currently receive imaging due to the contraindications of the conventional contrast agents. It avoids the use of ionizing radiation. Also, the conventional contrast agents are associated with risks. Iodinated contrast in CT is associated with significant risks of kidney damage. Another imaging technique, MR, uses gadolinium based contrast agents. Gadolinium, if used in patients with pre existing kidney dysfunction (defined as GFR < 30ml/min) is associated with the development of another devastating disease called nephrogenic systemic fibrosis. As HHT patients will require repeated scans throughout their lifetimes, this study will provide them a safer alternative.

Ten patients from the HHT clinic in whom the use of ferumoxytol as an MR agent is clinically indicated will be invited to participate in this study, which will determine if MR with ferumoxytol is able to detect and characterize vascular malformations in HHT.

DETAILED DESCRIPTION:
The safety of the use of gadolinium based contrast agents in MR is a concern for the FDA, with risks of development of nephrogenic systemic fibrosis and the more recent discovery of accumulation of gadolinium in the brain in patients who have received multiple prior MR scans.

Hereditary hemorrhagic telangiectasia (HHT) manifests with multiple vascular malformations (VMs) in the skin, mucous membranes and solid organs affecting the spine, brain, liver, gastrointestinal tract, pancreas, and lungs. The disease has an autosomal dominant inheritance and affects 1 in 5000 individuals.

Cerebral vascular malformations occur in 23 % of HHT patients, with a bleeding risk of 0.5% per year. Pulmonary AVMs occur in 15-50% of HHT patients, with a complication rate of 50% ranging from fatal hemoptysis or hemothorax to stroke or cerebral abscess. Liver vascular malformations are present in 32-78% of HHT patients.

The rationale for screening for vascular malformations is detection of a treatable lesion prior to the development of a fatal complication. The international guidelines currently recommend different first line screening tests in each organ: MRI for cerebral VMs, transthoracic echocardiography for pulmonary VMs, endoscopy for gastrointestinal VMs, Doppler US or CT for liver VMs.

Contrast enhanced magnetic resonance angiography (CE-MRA) may play an important role in the simultaneous whole body screening of vascular malformations. The advantages of CE-MRA include visualization of the entire body vasculature in one examination, high spatial resolution comparable to CT, no ionizing radiation and easy of multiplanar reconstructions.

Substituting a conventional gadolinium based contrast agent (GBCA) with an ultra small, super paramagnetic iron oxide agent (USPIO) e.g ferumoxytol, will eliminate any potential risk of developing nephrogenic systemic fibrosis. Since 2009, ferumoxytol ('Feraheme' Advanced Magnetics, Cambridge, MA) has been FDA approved for the treatment of iron deficiency anemia in adult patients with chronic kidney disease. The results of prior studies suggest that ferumoxytol is comparable to standard GBCAs for CE- MRA. Our experience with use of ferumoxytol to date suggests that it will be a superior agent for detection of vascular malformations in a range of vascular territories and that it will be uniquely capable of interrogating multiple territories in one sitting, due to its highly stable intravascular residence time.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of HHT (clinically or genetically confirmed)
* Known or suspected AVMs in the brain, lung, and/or liver
* Use of ferumoxytol as an MR agent is clinically indicated

Exclusion Criteria:

* Age <18
* Unable to have MRI scan
* Prior adverse reaction to ferumoxytol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Presence or absence of AVM | Immediate

SECONDARY OUTCOMES:
Size of AVM | Immediate
Location of AVM | Immediate
Overall image quality score | Immediate
Artifact score | Immediate
Vessel definition score | Immediate
Number of AVM feeding arteries | Immediate
Dimension of largest AVM feeding artery | Immediate
Number of AVM draining veins | Immediate
Dimension of largest AVM draining vein | Immediate
Dimension of aneurysmal sac | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Justin McWilliams, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No